CLINICAL TRIAL: NCT03917849
Title: Efficacy of Inertial Flywheel vs Heavy Slow Resistance Training Among Athletes With Patellar Tendinopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Nacional de Córdoba (Other)
Responsible Party: Principal Investigator, Diego Andres Ruffino, Principal Investigator, Universidad Nacional de Córdoba
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCordoba
Record Dates: First submitted 2019-04-08; First posted 2019-04-17 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Patellar Tendinitis; Jumper's Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Heavy slow resistance training (Experimental): The program is performed 3 times per week using resistance equipment in a fitness center. Each session consists of three 2-legged loaded quadriceps and lower limb kinetic chain exercises. The patients complete 3 or 4 sets in each exercise with a 2- to 3-minute rest between sets and a 5-minute rest period between the 3 exercises.
  The number of repetitions decreases, and load gradually increases, every week. The repetitions and loads are as follows: 3 times, 15-repetition maximum (15RM ), in week 1; 3 times, 12RM , in weeks 2 to 3; 4 times, 10RM , in weeks 4 to 5; 4 times, 8RM , in weeks 6 to 8; and 4 times, 6RM , in weeks 9 to 12.
  Interventions: Behavioral: Exercises program for patellar tendinopathy
- Inertial flywheel resistance training (Experimental): The program is performed 3 times per week using resistance equipment in a fitness center. Inertial flywheel resistance is a type of strength training; which is based on the increasing demands on eccentric action (breaking) after a concentric action (acceleration), due to the inertial load caused during the return movement. The patients complete 12 repetition máximum (RM) with moment inertia 0.05 m² from week 1-6 and 8 repetition máximum (RM) with moment inertia = 0.10 m² from week 6-12.
  Interventions: Behavioral: Exercises program for patellar tendinopathy

INTERVENTIONS:
Behavioral: Exercises program for patellar tendinopathy — To compare the effectiveness of the inertial flywheel resistance program versus slow heavy resistance in patients with chronic patellar tendinopathy

SUMMARY:
The purpose of this project is to investigate the efficacy of Inertial Flywheel Resistance program vs Heavy slow resistance in patients with chronic patellar tendinopathy.

The investigators hypothesize that Inertial Flywheel Resistance program will yield a more positive clinical outcome and function in patients with patellar tendinopathy compared to heavy slow resistance group.

DETAILED DESCRIPTION:
Randomized controlled intervention study

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of patellar tendinopathy
* Symptoms > 3 months
* Pain localized to the inferior pole of the patella
* Victorian Institute of Sport Assessment (VISA) score less than 80 points
* Palpation tenderness of the patellar tendon
* Abnormal tendon (hypoechoic) confirmed by ultrasonography.

Exclusion Criteria:

* Previous knee surgery
* Confounding diagnosis to the knee joint
* Previous corticosteroids injections
* Arthritis or diabetes

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Victorian Institute of Sports Assessment (VISA-P questionnaire) | 0 - 12 weeks
  Self-administered questionnaire. Consists of 8 items; 6 are used to evaluate pain levels or disability in daily activities and specific functional tests and 2 provide information regarding ability to play sport. Response options for each item are provided on a numeric rating scale (from 0 to 10), with higher scores indicating lower levels of pain or disability for all items other than 7 and 8, for which options have weighted scores.

SECONDARY OUTCOMES:
Patient-Specific Functional Scale | 0 - 12 weeks
  Self-reported patient-specific outcome measure assess functional change, primarily in patients presenting with musculoskeletal disorders. Patients are asked to identify up to 3 important activities they are unable to perform or are having difficulty with as a result of their problem. In addition to identifying the activities, patients are asked to rate, on an 11-point scale, the current level of difficulty associated with each activity. Following the intervention, patients are asked again to rate the activities previously identified.
Patient Global Impression of Change | 12 weeks
  Register patient's belief about the efficacy of treatment. PGIC is a 7 point scale depicting a patient's rating of overall improvement. Patients rate their change as "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Adverse events | 12 weeks
  To capture all adverse events and side effects that occurred after exercises protocol. Patients reported any changes or any symptoms. If a question was answered "yes", we asked for further comments.
Adherence self-report questionnaire | 12 weeks
  Patients were asked to choose one of six descriptions (from level 1 = perfect adherence to level 6 = nonadherence) to express exercise treatment at the end of the twelve weeks study period.
Single-leg decline squat (SLDS) test | 0 - 12 weeks
  A reliable patellar tendon pain provocation test, will be used to assess pain. Pain is rated on an 11-point numeric rating scale, where 0 is no pain and 10 is the worst pain imaginable.
Knee extension machine test | 0 - 12 weeks
  A reliable patellar tendon pain provocation test, will be used to assess pain. Pain is rated on an 11-point numeric rating scale, where 0 is no pain and 10 is the worst pain imaginable.
Jump test | 0 - 12 weeks
  Counter movement Jump and Triple hop for distance will be used to assess patellar tendinopathy caused functional deficits on the injured site compared with the non-injured site. The distance is measured in centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Vilma Campana, Dr, Study Director — Departments of Biomedical Physics - University of Cordoba Argentina
Locations (2):
- Argentina (2):
  - Universidad Nacional de Cordoba, Córdoba, C
  - Universidad Nacional de Cordoba, Córdoba

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruffino D, Malliaras P, Marchegiani S, Campana V. Inertial flywheel vs heavy slow resistance training among athletes with patellar tendinopathy: A randomised trial. Phys Ther Sport. 2021 Nov;52:30-37. doi: 10.1016/j.ptsp.2021.08.002. Epub 2021 Aug 4. PMID 34384941